CLINICAL TRIAL: NCT04687748
Title: Effects of Surface EMG-biofeedback on Pelvic Floor Muscle Training Among Women With Post-partum Urinary Incontinence.
Brief Title: EMG Biofeedback Based Pelvic Floor Training in Post Partum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/00836 Asma Jamshed
Record Dates: First submitted 2020-12-25; First posted 2020-12-29 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Urinary Incontinence
Keywords: Pelvic floor muscles; Electromyographic Biofeedback; pelvic floor strengthening
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: There will be two groups of participants, Experimental group will receive pelvic floor strengthening with EMGBF (Electromyographic Biofeedback ) and control group receive excercises without EMGBF.
Who Masked: Participant
Masking Description: Participants will be selected through purposive sampling technique per inclusion & exclusion criteria. Further, Randomization will be done by sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG BF Group (Experimental): Pelvic floor muscle contraction will be performed via an S-EMGBF device; patients in the s-EMGBF group will receive visual and auditory feedback.
  Interventions: Device: Electromographic Biofeedback
- Control Group (Active Comparator): Patients would be advised to maximally contract the pelvic floor muscles as forcefully a possible for about 5 seconds.
  Interventions: Other: PFM exercises

INTERVENTIONS:
Device: Electromographic Biofeedback — Surface EMG biofeedback is an adjunct therapy to standard exercise regime for increasing muscle strength. Electromyographic biofeedback is a specific form of biofeedback. The device records muscle activity through application of vaginal probe will be inserted in vagina and the reference surface electrode would be placed over the right anterior superior iliac spine.
  Arms: EMG BF Group
Other: PFM exercises — Patients would be advised to maximally contract the pelvic floor muscles as forcefully a possible for about 5 seconds. Three attempts would be made with 40 seconds rest in between each contraction. The exercises would be performed with the patient initially in supine position, with hip and knee flexed at 30 and 90 degrees.
  Arms: Control Group

SUMMARY:
This study intends to determine the effects of Electromyographic biofeedback on performance of pelvic floor muscles in urinary incontinence.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial ,will be conducted at Ripha Rehab Clinic,Rawalpindi. (EMG) biofeddback is a adjunct therapy to standard exercise regime for increasing muscle strength,this study is planned to determine the effects of electromyographic biofeedback on performance of pelvic floor muscles, strength,endurance ,rate of biofeedback and its impact on the qulatiy of life (QOL).The sample size was calculated to be n=28 through open-epitool version 3 ,with 95%confidence interval (CI),and power 80%.

After completion of therapeutic protocols, the participant will be assessed with the help EMG-biofeedback, Pelvic Floor distress inventory, King's Health Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Post-partum females
* Persistent urinary leakage at 3 months post-partum period
* Urine leakage with coughing, sneezing or exercise

Exclusion Criteria:

* Neurogenic bladder
* History of pelvic surgeries, pelvic tumors, UTI, urge incontinence, uncontrolled diabetes, cerebral stroke, previous injuries within pelvic

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Post partum females will be recruited in this study.
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle(PFM) Strength | Baseline
  To quantify PFM strength, the evaluator will insert the first two phalanges of the second and third fingers smeared in lubricant gel with a gloved hand into the anterior third of the vaginal opening and requested a maximal voluntary contraction by giving the command "squeeze my fingers". Muscle strength will be classified according to the modified Oxford scale into: 0 (nil), 1 (flicker), 2 (weak), 3 (moderate), 4 (good) to 5 (strong)
Pelvic floor muscle(PFM) Strength | Post 8th weeks
  To quantify PFM strength, the evaluator will insert the first two phalanges of the second and third fingers smeared in lubricant gel with a gloved hand into the anterior third of the vaginal opening and requested a maximal voluntary contraction by giving the command "squeeze my fingers". Muscle strength will be classified according to the modified Oxford scale into: 0 (nil), 1 (flicker), 2 (weak), 3 (moderate), 4 (good) to 5 (strong)
Pelvic distress inventory Questionnaire-20 | Baseline
  The PFDI-20 is comprised of 3 scales, which include the Urinary Distress Inventory-6 (UDI-6), Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory. The total score is out of 20.
Pelvic distress inventory Questionnaire-20 | post 8th week
  The PFDI-20 is comprised of 3 scales, which include the Urinary Distress Inventory-6 (UDI-6), Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory. The total score is out of 20.

SECONDARY OUTCOMES:
Kings health Questionnaire(KHQ) | Baseline
  Quality of life of patients will be measured by KHQ. It is a 10 items questionairre with rating on 4 item likert scale
Kings health Questionnaire(KHQ) | Post 8th weeks
  Quality of life of patients will be measured by KHQ. It is a 10 items questionairre with rating on 4 item likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Rehab Center RCRAHS Potohar campus, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nawaz H, Arshad H, Asim HM. Stress urinary incontinence after child birth - An unreported complication. J Pak Med Assoc. 2020 May;70(5):944. doi: 10.5455/JPMA.50445. No abstract available. PMID 32400762
- [Background] Anwer S QNMMEA. Effectiveness of electromyographic biofeedback training on quadriceps muscle strength in osteoarthritis of knee. 2011; 29(2)
- [Background] Kopanska M, Torices S, Czech J, Koziara W, Toborek M, Dobrek L. Urinary incontinence in women: biofeedback as an innovative treatment method. Ther Adv Urol. 2020 Jun 25;12:1756287220934359. doi: 10.1177/1756287220934359. eCollection 2020 Jan-Dec. PMID 32647538
- [Background] Chmielewska D, Stania M, Kucab-Klich K, Blaszczak E, Kwasna K, Smykla A, Hudziak D, Dolibog P. Electromyographic characteristics of pelvic floor muscles in women with stress urinary incontinence following sEMG-assisted biofeedback training and Pilates exercises. PLoS One. 2019 Dec 2;14(12):e0225647. doi: 10.1371/journal.pone.0225647. eCollection 2019. PMID 31790463
- [Background] Moroni RM, Magnani PS, Haddad JM, Castro Rde A, Brito LG. Conservative Treatment of Stress Urinary Incontinence: A Systematic Review with Meta-analysis of Randomized Controlled Trials. Rev Bras Ginecol Obstet. 2016 Feb;38(2):97-111. doi: 10.1055/s-0035-1571252. Epub 2016 Jan 29. PMID 26883864